CLINICAL TRIAL: NCT00515970
Title: Prospective Randomized Trial: Curettage Versus Excision in Nodular and Superficial Basal Cell Carcinomas
Brief Title: Curettage Versus Excision in Nodular and Superficial Basal Cell Carcinomas
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with the electronic data collection program
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Professor Helmut Breuninger, MD, Department of Dermatology, Eberhard Karls University, Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E.03.26007.1
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Carcinoma, Basal Cell
Keywords: Carcinoma, Basal Cell; Curettage; Excision; Recurrence; Complication; Esthetic outcome
MeSH Terms: conditions — Carcinoma, Basal Cell; Recurrence | interventions — Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Clinical or histologic diagnosis of nodular BCC
  Interventions: Procedure: Curettage
- 2 (Active Comparator): Clinical or histologic diagnosis of nodular BCC
  Interventions: Procedure: Deep excision
- 3 (Experimental): Clinical or histologic diagnosis of superficial BCC
  Interventions: Procedure: Curettage
- 4 (Active Comparator): Clinical or histologic diagnosis of superficial BCC
  Interventions: Procedure: Shave excision

INTERVENTIONS:
Procedure: Curettage — Curettage without subcutaneous tissue using a 7 mm ring curette and the "fountain-pen technique" (http://www.biopsypunch.com/kuerettagetechnik.htm; accessed on March 13, 2008). The curette is held between the thumb, index and middle finger. This method of holding enables precise guiding of the instrument, so that the piece of tissue can be removed in one well-targeted incision. After macroscopically complete removal, a safety margin is removed with the curette. It is used for histology to distinguish between R0 (excision margin without tumor cells) and R1 resection (excision margin containing tumor cells). Preparation with paraffin. Parallel, vertical sections for histologic diagnosis. Hematoxylin-eosin staining. Measurement of tumor thickness in mm.
  Arms: 1
Procedure: Deep excision — 12 o'clock mark. Excision with a scalpel down to the subcutaneous level. Plastic reconstruction. Three vertical, parallel bread loaf sections for histology. Preparation with paraffin. Staining with hematoxylin-eosin. Histologic diagnosis including report of tumor thickness in mm. Comment on complete removal (R0 versus R1). In case of R1 excision directed reoperations are performed until R0 is achieved.
  Arms: 2
Procedure: Shave excision — Shave excision with a safety margin, using a scalpel. Wound healing by secondary intention. Preparation with paraffin. Parallel vertical bread loaf sections for histology. Staining with hematoxylin-eosin. Histologic diagnosis. Comment on complete removal (R0 versus R1). In case of R1 excision a reoperation is performed until R0 is achieved.
  Arms: 4
Procedure: Curettage — Curettage with a 7 mm ring curette with the "potato-peeler technique" (http://www.biopsypunch.com/kuerettagetechnik.htm; accessed on March 13, 2008). The handle of the curette is held in the distal inter-digital fold of the index finger, and supported by the other fingers of the curetting hand. The thumbs serve to provide a stable base. This technique makes it possible to guide the instrument, applying greater pressure, but accuracy is reduced. After macroscopically complete removal, a safety margin is removed with the curette. It is used for histology to distinguish between R0 (excision margin without tumor cells) and R1 resection (excision margin containing tumor cells). Preparation with paraffin. Parallel, vertical sections for histologic diagnosis. Hematoxylin-eosin staining.
  Arms: 3

SUMMARY:
Basal cell carcinoma (BCC) is the most frequent skin cancer. Uncontrolled growth destroys local anatomic structures. There are various treatment alternatives with different recurrence rates and expenses. After surgical excision, the recurrence rate is in between 3 and 4% and the procedure is relatively expensive. Photodynamic therapy as well as imiquimod 5% are expensive therapies with high recurrence rates, that lack histologic evidence of BCC. Cryosurgery and curettage are inexpensive, although the recurrence rates are higher than after surgical excision.

This prospective, randomized trial compares recurrence rates, cosmetic outcome, and surgery-related complications after curettage versus surgical excision in nodular and superficial BCC. About 600 tumors will be included. One half is treated by curettage, the other half by surgical excision. The follow-up period is four years. If the difference between recurrence rates is ≤7% and the cosmetic outcome as well as the surgery-related complications are not worse after curettage, surgical excision must be considered an overtreatment.

DETAILED DESCRIPTION:
1. First presentation of a patient with clinical or histopathological diagnosis of BCC
2. Study patient number, first and surname, date of birth and gender are listed in a distinct file.
3. Informed consent
4. Whole body screening for skin cancer
5. In- or exclusion of the patient. If the patient is excluded, no more data are obtained.
6. Recording of the following features in an electronic file:

   1. Number of BCCs
   2. Anatomic location

      * Lip
      * Eyelid
      * Ear
      * Nose
      * Other parts of the face
      * Scalp or neck
      * Trunk
      * Arm, hand, or shoulder
      * Leg, foot, or hip
   3. Position

      * Ventral or dorsal. If the tumor is located at the lateral margin of ventral and dorsal, it is considered ventral.
      * Right, left, midline
      * Distinct BCCs are numbered. To ensure future distinction of different tumors, numbering starts with the most up-right-ventral tumor and ends with the most down-left-dorsal one. Numbering continues with BCCs that appear later during the period of recruitment.
   4. Diameter in mm
7. In- or exclusion of the tumor
8. Photographs of the included BCCs
9. Randomization is performed by the Department of Biostatistics (distance to the Department of Dermatology = 1.7 km) with envelopes containing the assigned study arm. The study physician calls one of four staff members of the Department of Biostatistics and asks for randomization. The envelopes are not opened unless the electronic data file is completed by the study physician.
10. Disinfection
11. Local anesthesia
12. Surgery
13. Dressing
14. If histopathology discovers another BCC type than nodular or superficial or even another tumor than BCC, then the tumor is excluded.
15. Follow-up visit 3 and 6 months (+/- 30 days) after the operation. In BCCs that had to be operated in >1 step, the day of the follow-up visit refers to the initial operation.
16. In case of clinical suspicion of recurrence of BCC a punch biopsy is taken. If the biopsy confirms recurrence, the endpoint is achieved.
17. If BCCs must be added to a patient during the recruitment period, follow-up visits always refer to the latest BCC.
18. If the patient visits our department not within the defined follow-up period, the appointment is not recorded (except confirmation of recurrence).
19. Patients who provide no feedback receive phone calls.
20. If a patient or a private practitioner suspect a recurrence of BCC beyond a defined follow-up period, of course, the patient is invited as early as possible to our department, where a biopsy will be taken.
21. The patient receives a letter containing a list of the BCCs treated within the study. The private practitioner is to be visited with the list after 12, 24, and 36 months (+/- 30 days) referring to the last operation within the recruitment period. The letter contains a questionnaire about scar size and suspicion of recurrence of BCC. The practitioner or the patient return the questionnaire with the answers to our department. If recurrence is suspected we take a biopsy.
22. When follow-up is closed for an individual patient, the reason is recorded:

    1. Planned end of follow-up after 48 months.
    2. Patient has moved.
    3. Death (date of death).
    4. Consent withdrawn.
    5. Patient has become meanwhile so ill or high-maintenance that no more follow-up visits can be planned.
    6. Recurrence of all of the patient's BCCs.
23. Statistic evaluation is based on an intention-to-treat-analysis.
24. The trial is designed to prove the equivalence of treatment modalities. A statistic test is used for evaluation, including the Kaplan-Meier-method. When all 4 study arms contain 116 BCCs, a 2-group-test on the equivalence of ratios with a 1-sided significance level of 0.05 will have a power of 80% to disprove the null hypothesis. The null hypothesis is that standard and test method are not equivalent (ratio difference delta T - delta S ≥ 0.15). Then the alternative hypothesis is more probable, meaning that the ratios in both groups are equivalent supposed that the expected ratio difference is 0.07 and the ratio within the standard group is 0.03 (according to an expected recurrence rate of 3% in the surgical excision study arm).

ELIGIBILITY:
Inclusion Criteria:

* Clinical or histologic diagnosis of BCC

Patient Dependent Exclusion Criteria:

* > 5 BCCs at presentation
* Immunosuppressive drugs
* Pregnancy
* Disability to give informed consent
* Synchronous participation in other studies
* Progeroid syndromes
* Other malignant tumors, except for BCC and squamous cell carcinoma, or monoclonal neoplasms of the hematopoietic or immune system
* Critical illness precluding sufficient follow-up visits

Tumor Exclusion Criteria:

* Recurrent BCC
* Nodular BCC with an exophytic part of > 1.5 mm above skin level
* Nodular BCC with a diameter of > 10 mm
* Superficial BCC with a diameter of > 20 mm
* Ulceration
* Scarring
* Blurred margins
* Histopathologic evidence of a tumor type different from nodular or superficial BCC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of BCC, confirmed by biopsy | 4 years after surgery

SECONDARY OUTCOMES:
Secondary hemorrhage as remembered by the patient | 3 months (plus or minus 30 days) after surgery
Wound infection as remembered by the patient | 3 months (plus or minus 30 days) after surgery
Hypesthesia after surgery | 3 months (plus or minus 30 days) after surgery
Keloid | 3 months (plus or minus 30 days) after surgery
Functional impairment or disfigurement by the scar. Keloid is always a disfiguring scar. If the scar is recognized as keloid, the measure "disfigurement" cannot be used here. | 3 months (plus or minus 30 days) after surgery
Subjective assessment of the esthetic outcome of the scar on a scale of excellent, good, satisfying, moderate, unfavorable; done by the patient | 3, 6, 12, 24, 36, and 48 months (plus or minus 30 days) after surgery
Subjective assessment of the esthetic outcome of the scar on a scale of excellent, good, satisfying, moderate, unfavorable; done by the study physician | 3, 6, 12, and 48 months (plus or minus 30 days) after surgery
Subjective assessment of the esthetic outcome of the scar on a scale of excellent, good, satisfying, moderate, unfavorable; done by a private practitioner | 12, 24, and 36 months (plus or minus 30 days) after surgery
Scar length in mm | 6 and 48 months (plus or minus 30 days) after surgery
Scar width in mm, perpendicular to its length | 6 and 48 months (plus or minus 30 days) after surgery
Color of the scar: hyperpigmented, hypopigmented, or erythematous | 6 and 48 months (plus or minus 30 days) after surgery
Level of the scar: atrophic, skin level, hypertrophic, or keloid | 6 and 48 months (plus or minus 30 days) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Breuninger, M.D., Study Chair — Department of Dermatology, Eberhard Karls University Tuebingen
Locations (1):
- Department of Dermatology, Eberhard Karls University, Tübingen, Baden-Wurttemberg, Germany